CLINICAL TRIAL: NCT06254092
Title: Effect of Tourniquet Binding of Cervical on the Blood Volume of Amniotic Fluid in Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, zhiming zhang, chief, First People's Hospital of Chenzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023121
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Amniotic Fluid Embolism; Pulmonary Hypertension
Keywords: amniotic fluid entering the bloodstream; blood volume of amniotic fluid; Amniotic fluid embolism
MeSH Terms: conditions — Embolism, Amniotic Fluid; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tourniquet (Experimental): The investigators use tourniquets to bind the cervical for intervention groups to block venous return to the lower uterine segments to reduce the inflow of amniotic fluid into the uterus.
  Interventions: Procedure: tourniquet binding of cervical

INTERVENTIONS:
Procedure: tourniquet binding of cervical — The procedure will be performed by surgeons with rich experience in clinical work

SUMMARY:
This study was conducted to investigate whether the use of tourniquet after delivery of the fetus could reduce the amount of amniotic fluid entering the bloodstream and thus reduce the incidence of intraoperative adverse events.

DETAILED DESCRIPTION:
Amniotic fluid embolism (AFE) is a rare complication specially to obstetrics.When amniotic fluid enters the maternal circulation , a sudden onset of a series of pathophysiologic changes such as pulmonary hypertension, hypoxemia, circulatory failure, disseminated intravascular coagulation, and multiorgan failure may occur. Routinely, the typical AFE triad is uneasy to discover, and nonspecific adverse reactions such as irritability, chills, chest tightness and shortness of breath, transient drop in blood pressure, and nausea and vomiting are often seen during delivery of the fetus and placenta. All of the above symptoms may suggest that the amniotic fluid has entered into the bloodstream. In clinical anesthesia, investigators observed that women with placenta praevia and placenta implantation were less likely to suffer these nonspecific symptoms after delivery of the fetus compared with women with normal pregnancies.The investigators speculated it might be related to the fact that obstetricians used tourniquets to reduce intraoperative hemorrhage in the former, blocking venous return to the lower uterine segments to reduce the inflow of amniotic fluid into the uterus. Therefore, this study was conducted to investigate whether the use of tourniquet after delivery of the fetus could reduce the amount of amniotic fluid entering the bloodstream and thus reduce the incidence of intraoperative adverse events.

ELIGIBILITY:
Inclusion criteria

1. Single pregnancy
2. Be in good health, with no high blood pressure or heart disease during pregnancy
3. Without placenta previa and placenta implantation
4. No abdominal adhesions, suitable for operation
5. Signed informed consent by the pregnant woman and her family

Exclusion criteria

1. Serious coagulation abnormality
2. Preoperative severe cardiac, cerebral, pulmonary, hepatic, renal and other important organs insufficiency and electrolyte abnormality combined with placenta praevia or placenta implantation
3. Multiple pregnancies
4. Previous history of abdominal surgery
5. Intraoperative drug allergy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
sTn | before the fetus is delivered,after the fetus is delivered,before the puerpera is sent back to the ward
  sTn refers to meconium and mucin extracted from amniotic fluid. The presence of sTn in the patient's serum is a diagnostic method that can directly prove that mucin derived from amniotic fluid has entered the maternal circulation.

SECONDARY OUTCOMES:
HR MAP | before the fetus is delivered,after the fetus is delivered,before the placenta is delivered,after the placenta is delivered,after releasing the tourniquet,before the puerpera is sent back to the ward
  Measurement of HR by patient monitor and MAP by placing an arterial puncture catheterization.
SPO2,PaO2,PaCO2 | before the fetus is delivered,after the fetus is delivered,before the placenta is delivered,after the placenta is delivered,after releasing the tourniquet,before the puerpera is sent back to the ward
  the respiratory parameters in arterial blood gas
Thrombelastogram(TEG) | before the fetus is delivered,before the puerpera is sent back to the ward
  Thrombelastography (TEG) is an indicator of the dynamic changes of blood coagulation. It can evaluate thrombelastography and compensate for the failure of routine examinations to reflect the fibrinolytic system and platelet function.
Adverse events | perioperatively
  Irritability, chills, chest tightness and shortness of breath, transient drop in blood pressure, and nausea and vomiting
Hemorrhage | before the puerpera is sent back to the ward, 2 hours after the puerpera back to ward
  The using of tourniquets can reduce intraoperative hemorrhage. The postpartum hemorrhage reflects the coagulation function of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming zhang, Principal Investigator — Chenzhou NO. 1 people's Hospital
Locations (1):
- Zhiming Zhang, Chenzhou, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided